CLINICAL TRIAL: NCT06851949
Title: Vsling™ I: Clinical Evaluation of the Vsling™ Device for Ventricular Repair in Patients With Heart Failure
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cardiac Success (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-9003
Record Dates: First submitted 2025-01-01; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Vsling (Experimental): Vsling Device implantation
  Interventions: Device: Vsling

INTERVENTIONS:
Device: Vsling — Implantable ventricular repair device

SUMMARY:
Prospective, multi-center, open-label clinical study of the feasibility and initial safety and performance of the Vsling™ in patients with heart failure (HF) with evidence of reduced left ventricular ejection fraction, associated with ventricular dilation.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years
2. Left ventricular end diastolic diameter is greater than or equal to 55mm
3. Ejection fraction ≥20% and ≤40%
4. FMR grade ≤ 2+ (≤ mild FMR) as defined by the guidelines of the American society of echocardiography (via a transthoracic or transesophageal echo)
5. End-systolic Interpapillary muscle distance ≥ 20mm
6. NYHA class II-IVa
7. Cardiomyopathy of ischemic or non-ischemic origins
8. Understands the nature of the study and procedure and able to provide written informed consent

Exclusion Criteria:

1. Any evidence of structural (chordal or leaflet) mitral lesions
2. Ventricular tachycardia or ventricular fibrillation within 6 months prior to inclusion in this study
3. Prior mitral valve repair or replacement
4. ICD/CRT/cardiac pacemaker leads implanted within 3 months prior to inclusion in this study
5. Clinical signs of cardiogenic shock within 30 days prior to inclusion in this study
6. Anatomy that, in the opinion of the interventionalist, prevents safe passage of the Vsling™ catheter(s).
7. Severe aortic stenosis
8. Severe, massive, or torrential tricuspid regurgitation requiring surgical or transcatheter repair
9. Known fixed pulmonary hypertension with PA systolic pressure >70 mmHg not responsive to vasodilator therapy
10. ST segment elevation myocardial infarction within 30 days prior to inclusion in this study
11. Congenital heart disease (except PFO, PDA or ASD)
12. Heart Failure due to confirmed amyloid or other restrictive cardiomyopathies
13. Chronic renal insufficiency defined by Creatinine ≥ 3.0 mg/dL or chronic renal replacement therapy
14. Any therapeutic invasive cardiac procedure within 30 days prior to index procedure
15. Any cardiac surgery, within 3 months prior to inclusion in the study
16. Cerebrovascular Accident (CVA) within 90 days prior to inclusion in this study
17. Thrombocytopenia (Platelet count< 100,000/mm3) or thrombocytosis (Platelet count > 750,000/mm3)
18. Body temperature >38°C within 3 days prior to index procedure
19. Bleeding disorders or hypercoagulable state
20. Active peptic ulcer or active gastrointestinal (GI) bleeding within 90 days of the scheduled implant
21. Contraindication to anticoagulants or antiplatelet agents
22. Known allergy to stainless steel, nickel, titanium or contrast agents that cannot be adequately pre-medicated
23. Known hypersensitivity or contraindication to procedural medications which cannot be adequately managed medically
24. Currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study
25. Co-morbid condition(s) that, in the opinion of the Investigator, limit life expectancy to < 12 months
26. Co-morbid condition(s) that, in the opinion of the investigator, could limit the patient's ability to participate in the study, including compliance with follow-up requirements, or that could impact the scientific integrity of the study
27. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Device related Serious Adverse Events (SAE) | 30 Days
  Device related Serious Adverse Events (SAE) within 30 days of the procedure: any SAE that has been determined by the safety monitor to be related to the Vsling™ implantation procedure or the Vsling™ device

CONTACTS AND LOCATIONS:
Locations (5):
- Israel (5):
  - Shamir Medical Center, Be’er Ya‘aqov
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Tzafon Medical Center, Poria – Neve Oved

IPD SHARING:
Plan to Share IPD: Undecided